CLINICAL TRIAL: NCT04762927
Title: Metric Properties of de Morton Mobility Index in Rehabilitation Patients With Musculoskeletal Impairments
Brief Title: Metric Properties of de Morton Mobility Index
Acronym: DEMMIURIS
Status: Completed | Type: Observational
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Other Study IDs: URIS202101
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Musculoskeletal Diseases
Keywords: DEMMI; outcome measurement; physiotherapy; clinimetric properties
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metric properties (convergent validity, predict validity, known-groups validity, responsiveness, floor and ceiling effects, minimal clinically important difference) of the de Morton Mobility Index (DEMMI) in patients with musculoskeletal impairments undergoing impatient rehabilitation will be investigated.

DETAILED DESCRIPTION:
Convergent validity of DEMMI will be assessed in terms of correlations with the other outcome measures. Known-groups validity will be demonstrated by differences in DEMMI scores between patients who were not able to walk and those who were able to walk with or without walking aid. Predictive validity of DEMMI at admission for functional independence at discharge from rehabilitation will be estimated. The minimal clinically important difference of DEMMI, responsiveness and floor or ceiling effects will also be estimated.

ELIGIBILITY:
Inclusion Criteria:

* admission to inpatient rehabilitation
* written informed consent

Exclusion Criteria:

* associated impairments of the central nervous system or other severe health conditions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with musculoskeletal impairments with or without impairments of peripheral nerves
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
de Morton Mobility Index - change | Approximately 30 days (difference between admission and discharge)
  DEMMI is a unidimensional 15-item measure of mobility for adults

SECONDARY OUTCOMES:
Ten-meter Walk Test | Approximately 30 days (difference between admission and discharge)
  10mWT assesses comfortable walking speed over the distance of 10 meters
Six-minute Walk Test - change | Approximately 30 days (difference between admission and discharge)
  6mWT assesses assess aerobic capacity and endurance
Functional Independence Measure - change | Approximately 30 days (difference between admission and discharge)
  FIM is an 18-item two-dimensional instrument that explores physical and psychosocial functioning
EQ-5D-3L - change | Approximately 30 days (difference between admission and discharge)
  EQ-5D-3L is a patient-reported instrument for measuring HRQOL

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Zupanc, PT, MSc, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia